CLINICAL TRIAL: NCT04547452
Title: Combination of Sintilimab and Stereotactic Body Radiotherapy in Advanced Metastatic Hepatocellular Carcinoma
Brief Title: Combination of Sintilimab and Stereotactic Body Radiotherapy in Advanced Metastatic HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Wang Xin, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-SBRT-HCC-001
Record Dates: First submitted 2020-09-06; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-07

CONDITIONS: Stage IV HCC; Immunotherapy; SBRT
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab Combined with SBRT (Experimental): Patients will be randomly placed in either of the two arms. Participants enrolled in this arm treated to a total dose of 35-80Gy in 5-8 fractions with stereotactic radiotherapy to a liver or lung or any metastatic lesion. The choice of radiation dose will be at the discretion of the treating radiation oncologist.
  Sintilimab is administered intravenously at 200 mg every 3 weeks for up to 1 year.
  Interventions: Radiation: Stereotactic body radiation therapy; Drug: Anti-PD-1 antibody drug named Sintilimab
- Sintilimab (Active Comparator): Participants enrolled in this arm treated with sintilimab administered intravenously at 200 mg every 3 weeks for up to 1 year.
  Interventions: Drug: Anti-PD-1 antibody drug named Sintilimab

INTERVENTIONS:
Radiation: Stereotactic body radiation therapy — Sintilimab Combined with SBRT
  Other Names: SBRT
  Arms: Sintilimab Combined with SBRT
Drug: Anti-PD-1 antibody drug named Sintilimab — Sintilimab

SUMMARY:
Hepatocellular carcinoma (HCC) is a common malignancy, and more than 70% of newly diagnosed HCC patients already have advanced disease. Sorafenib and lenvatinib are recommended as first-line options for advanced HCC. The PD-1 monoclonal antibody，such as nivolumab and pembrolizumab, have been approved to treat the patients with advanced HCC by the FDA. Combining radiotherapy with immune checkpoints showed promising response rates and improved survival in several solid tumor types. The purpose of this randomized study is to determine whether stereotactic body radiation therapy (SBRT) combined with sintilimab (an anti-PD-1 antibody) will improve the response to the anticancer treatment compared to sintilimab alone in patients with advanced HCC.

About 84 participants will be enrolled in this study. All will take part at West China Hospital, Sichuan University.

DETAILED DESCRIPTION:
A total of 84 HCC patients who are failure from the first line Sorafenib or lenvatinib treatment will be randomized to two treatment arms using a 1:1 ratio: SBRT + PD-1 arm or PD-1 alone arm.

Patients in both arms will receive sintilimab administered intravenously at 200 mg every 3 weeks. Stereotactic body radiotherapy (SBRT) using volumetric arc therapy. The prescribed dose is 30-54 Gy in 3-6 fractions over 1-2 weeks. In the SBRT + PD-1 arm, sintilimab is administered intravenously at 200 mg every 3 weeks for up to 1 year. The first course of sintilimab will be given within 4-6 weeks after completion of SBRT.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed hepatocellular carcinoma or diagnosed by American Association for the Study of Liver Disease criteria;
2. Deemed ineligible for curative intent therapy with surgical resection or liver transplantation.
3. Estimated life expectancy ≥12 weeks;
4. Male or female subjects with age: 18-70 years old
5. Failure in first-line systemic treatment with sorafenib or Lenvatinib
6. Unwilling to receive or unable to tolerate first-line treatment with sorafenib
7. Have ECOG performance status 0-1
8. Have measurable disease based on RECIST 1.1.
9. Pretreatment CT chest /abdomen /pelvis within 28 days of protocol enrollment.
10. Child-Pugh class A liver function (assessed within 14 days of SBRT)；
11. The function of important organs meets the following requirements: a. white blood cell count (WBC) ≥ 3.0×109/L, absolute neutrophil count (ANC) ≥ 1.5×109/L; b. platelets ≥ 50×109/L; c. hemoglobin ≥ 8g/dL; d. serum albumin ≥ 3.0g/dL; e. total bilirubin ≤ 2.0×ULN, ALT, AST ≤ 5×ULN; f. serum creatinine ≤ 1.5×ULN
12. Must have at least one lesion amenable to SBRT.
13. Ability to understand the study and sign informed consent.

Exclusion Criteria:

1. A history of abdominal radiotherapy;
2. Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (positive for hepatitis C antibody, and HCV-RNA levels higher than the lower limit of the assay);
3. Active autoimmune diseases, a history of autoimmune diseases (including but not limited to these diseases or syndromes, such as colitis, hepatitis, hyperthyroidism), a history of immunodeficiency (including a positive HIV test result)
4. History of organ transplantation or allogeneic bone marrow transplantation，or other acquired or congenital immunodeficiency diseases
5. Receipt of live, attenuated vaccine within 30 days prior to the study treatment
6. Has a known history of active TB (Bacillus Tuberculosis).
7. Uncontrolled intercurrent illness including, but not limited to digestive tract ulcer, uncontrolled hypertension, fracture, uncured wound, history of congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
8. Prior invasive malignancy within 2 years except for noninvasive malignancies such as cervical carcinoma in situ, in situ prostate cancer, non-melanomatous carcinoma of the skin, lobular or ductal carcinoma in situ of the breast that has been surgically cured
9. Female patients who are pregnant or lactating
10. Untreated central nervous system (CNS) metastatic disease, lepto-meningeal disease, or cord compression
11. Active infection requiring systemic therapy
12. Presence of clinically meaningful ascites，hydrothorax or hydropericardium and patients requiring non pharmacologic intervention (eg, paracentesis) or escalation in pharmacologic intervention to maintain symptomatic control
13. Severe hypersensitivity reaction to treatment with another monoclonal antibody (mAb)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
24-week progression-free survival (PFS) ratev | 24 weeks after radiotherapy
  The proportion of patients with progression disease according to mRECIST at 24 weeks from randomization.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months after the enrollment
  Investigator assessed ORR using RECIST v1.1 including the all tumor, the tumor undergoing LDRT and the tumor which do not receive radiotherapy.
Overall Survival (OS) | up to 24 months after the enrollment
  OS is defined as the difference (in months) between the date of study enrollment to the date death due to any cause
24-week disease control rate (DCR) | 24 weeks after radiotherapy
  The proportion of patients with complete response, partial response or stable disease according to mRECIST at 24 weeks from randomization.
Duration of response (DOR) | up to 24 months after the enrollment
  From date of first CR/PR to the date of first PD according to RECIST criteria, assessed up to 24 months.
Adverse Events | 2 years from randomization
  Treatment-related adverse events are graded according to the Common Toxicity Criteria, version 4.0, and were registered from the date of informed consent until discontinuation of trial treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No